CLINICAL TRIAL: NCT02947490
Title: Trial of the Effectiveness and Cost Effectiveness of Self-monitoring and Treatment of Blood Pressure in Secondary Prevention Following Stroke or Transient Ischaemic Attack (TIA)
Brief Title: Effectiveness of Self-monitoring and Treatment of Blood Pressure Following Stroke or Transient Ischaemic Attack
Acronym: TEST-BP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JPotter
Record Dates: First submitted 2015-05-21; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
Keywords: Blood pressure monitoring; self BP monitoring; self BP management
MeSH Terms: conditions — Stroke | interventions — Standard of Care; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard BP management (Sham Comparator): Participants will continue to receive routine measurement of BP and management of treatment from their General Practitioner (GP).
  Interventions: Other: Standard BP management
- Self BP measurement and standard care (Placebo Comparator): Participants in this group (Se-Mo) will be taught to use a validated British Hypertension Society (BHS) approved home BP monitor (with built in memory/printer) by the study nurse along with written information on the procedure and a copy of the BHS Home BP Monitoring DVD. Participants will be contacted before each recording week & arrangements will be made to deliver and demonstrate the use of self BP monitor by the study nurse. Home BP monitoring will be performed over a 7 day period 3 times during the 6 month follow-up and on each occasion the patient will be given a copy of the BP results and asked to inform the GP of the results and the GP will decide if any alteration in therapy is needed.
  Interventions: Other: Self BP measurement; Other: Standard Care
- Self BP measurement and treatment (Active Comparator): Participants in this group will undergo exactly the same self BP monitoring training process as the Se-MO group and will undertake monitoring at the same time intervals. However they will be equipped with a validated BP monitor with a Bluetooth interface phone, BP values recorded by the patient will be transmitted automatically via mobile telephone to the trial coordinating centre. The data will be password protected and saved on a secure server and be available only to the trial team (study nurse & supervising physicians). The patient would then be contacted by the study nurse and depending on BP levels recorded the patient will alter their medication to achieve target BP levels. This will be recorded on the CRF and the GP notified of any treatment changes.
  Interventions: Other: Standard Care; Other: Treatment

INTERVENTIONS:
Other: Self BP measurement — BP home measurement by patient, results to GP and GP alters treatment as per usual practice
  Arms: Self BP measurement and standard care
Other: Standard Care — Self BP measurement and patient management of anti-hypertensive treatment altering their own medication under supervision depending on home BP measurements
  Arms: Self BP measurement and standard care; Self BP measurement and treatment
Other: Standard BP management — GP to measure BP and manage BP control
  Arms: Standard BP management
Other: Treatment — Contacted by the study nurse and depending on BP levels recorded the patient will alter their medication to achieve target BP levels.
  Arms: Self BP measurement and treatment

SUMMARY:
This blinded end point RCT will recruit high risk TIA and mild stroke patients (through the emergency TIA clinics and the acute stroke services at the Norfolk & Norwich University Hospital) who require anti-hypertensive therapy to examine the clinical and cost effectiveness of self-monitoring and self management of Blood Pressure compared to self monitoring alone and treatment as usual.

DETAILED DESCRIPTION:
Research Question: In patients with a mild/moderate stroke or TIA who require drug treatment for BP control, does BP self-monitoring with or without patient-led management using a previously agreed treatment regime result in better BP control and patient satisfaction than standard GP based management?

Planned sample size: 165 eligible participants distributed 1:1:1 between three groups. Group 1 (control) - treatment as usual (TAU). Group 2 - Self-monitoring only (Se-MO). Group 3 - Self-monitoring and self-management (Se-Man).

Primary outcome: Number reaching target Ambulatory BP levels at follow-up and change in mean Ambulatory BP levels between baseline and follow-up at 6 months.

Secondary outcomes:

Number of changes in anti-hypertensive treatment during study Side-effects profiles and adverse events BP variability Pulse Wave Velocity (PWV) changes All cause and cause-specific mortality outcome at six month Recurrent TIA or stroke Incident CVD- stroke, TIA and myocardial infarction Costs Health related quality of life assessed Quality Adjusted Life Years (EQ-5D based) Patient satisfaction and experience of the process (qualitative data)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged =/> 18 years old with TIA or stroke of mild/moderate severity (NIHSS =<15) who require BP management and are able and willing to undertake self BP measurement and guided alterations in therapy.

Exclusion Criteria:

* Those with terminal illness with life expectancy less than six months including end staged condition e.g. end stage COPD
* Dementia or moderate to severe cognitive impairment
* Those not receiving or expected to start anti-hypertensive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2013-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in mean daytime/24 hour BP between baseline and follow-up using 24 hour BP recording and numbers reaching target BP | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Potter, DM FRCP, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided